CLINICAL TRIAL: NCT02498015
Title: A Phase IV Open-label, Multicentre, International Trial of Paritaprevir/Ritonavir, Ombitasvir, Dasabuvir ±Ribavirin for Chronic Hepatitis C Virus Genotype 1 Infection and Recent Injection Drug Use or Receiving Opioid Substitution Therapy
Brief Title: A Phase IV Trial of Paritaprevir/Ritonavir, Ombitasvir, Dasabuvir for Chronic Hepatitis C Genotype 1 Virus Infection
Acronym: D3FEAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1405
Record Dates: First submitted 2015-06-26; First posted 2015-07-15 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "3D" regimen (Experimental): The "3D" regimen contain two tablets of co-formulated paritepravir/ritonavir/ombitasvir (75/50/12.5 mg) once daily, and one dasabuvir tablet (250 mg) twice daily for genotype 1b without cirrhosis. Treatment will be 12 weeks.
  Interventions: Drug: "3D" regimen
- "3D" regimen with ribavirin (Experimental): The "3D" regimen with ribavirin contain two tablets of co-formulated paritepravir/ritonavir/ombitasvir (75/50/12.5 mg) once daily, one dasabuvir tablet (250 mg) twice daily, and ribavirin (1000 mg regardless of weight) daily in two divided doses for genotype 1a (with/without) and genotype 1b with cirrhosis. Treatment will be for 12 weeks.
  Interventions: Drug: "3D" regimen with ribavirin

INTERVENTIONS:
Drug: "3D" regimen — The "3D" regimen contain paritaprevir/ritonavir/ombitasvir (75/50/12.5mg) once daily, dasabuvir 250mg twice daily for genotype 1b without cirrhosis.
  Other Names: Viekira pack
  Arms: "3D" regimen
Drug: "3D" regimen with ribavirin — The "3D" regimen with ribavirin contain paritaprevir/ritonavir/ombitasvir (75/50/12.5mg) once daily, dasabuvir 250mg twice daily, and ribavirin (1000 mg regardless of weight) daily in two divided doses for genotype 1a and genotype 1b with cirrhosis.
  Other Names: Viekira pack with ribavirin
  Arms: "3D" regimen with ribavirin

SUMMARY:
A total of 100 people with chronic HCV and recent injection drug use or recipients of opioid substitution therapy will be enrolled in 5 countries and 21 study sites. Participants with genotype 1a infection or cirrhosis will receive 12 weeks of open-label paritaprevir/ritonavir/ombitasvir and dasabuvir ("3D"), and twice-daily ribavirin. Participants with genotype 1b infection without cirrhosis will receive 12 weeks of open-label "3D". The study consists of a screening phase (6 weeks), treatment phase (12 weeks) and follow-up phase (96 weeks) to evaluate treatment response and reinfection.

DETAILED DESCRIPTION:
A total of 100 people with recent injection drug use or recipients of opioid substitution therapy will be enrolled from drug and alcohol clinics, tertiary liver and infectious diseases clinics and community health centres across Canada, Europe, New Zealand, France, and Australia. This will include at least 30 participants with F3/F4 liver disease. Participants will be considered recent injection drug users if they have used injection drugs in the 6 months prior to consent. Participants receiving stable opioid substitution therapy (stable dose for >2 weeks) will also be included. Patients with frequent drug use that is judged by the treating physician to compromise treatment safety will be excluded. The study drugs consisting of two tablets of the co-formulated paritepravir/ritonavir/ombitasvir (75/50/12.5 mg) once daily, one dasabuvir tablet (250 mg) twice daily, ribavirin (1000 mg) daily in two divided doses (genotype 1a only and/or cirrhosis). Electronic blister packs will be used to improve and monitor treatment adherence. This innovative strategy with the "3D" interferon-free regimen could considerably enhance the capacity to scale-up HCV treatment among PWID, and is therefore being evaluated in this phase IV study within a well-defined PWID population.

ELIGIBILITY:
Inclusion criteria:

1. Detectable HCV RNA in plasma (>1,000 IU/ml).
2. Evidence of positive HCV antibody >6 months prior to screening.
3. HCV Genotype 1 infection.
4. Recent IDU (previous 6 months) or receiving stable OST (stable dose for >2 weeks).
5. Never received treatment for HCV infection.
6. Compensated liver disease. Enrolment of patients with cirrhosis (FibroScan >14.6 kPa or FIB-4 > 3.25) will be capped to 60% of the total enrolment (maximum 3 per site).
7. Participants with FibroScan > 12KPa or AFP >50 ng/mL must have abdominal ultrasound or CT scan without evidence of hepatocellular carcinoma within 2 months before screening.
8. Negative pregnancy test (for women of childbearing potential) within the 24-hour period before the first dose of study drug.
9. All fertile participants must be using effective contraception during treatment and 24 weeks post treatment (patients treated with ribavirin) or 2 weeks post treatment (patients not treated with ribavirin).

Exclusion criteria:

1. Any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) ≤6 months before the first dose of study drug.
2. Any investigational drug ≤6 weeks before the first dose of study drug.
3. HIV infection.
4. History or other evidence of decompensated liver disease.
5. Neutrophil <1000 cells/mm3 or platelet <50,000 cells/mm3 at screening.
6. Serum creatinine >1.5 x upper limit of normal at screening.
7. Ongoing severe psychiatric disease as judged by the treating physician.
8. Frequent IDU that is judged by the treating physician to compromise treatment safety.
9. Hemoglobin <12 g/dL (<7.4 mmol/L) in women or <13 g/dL (<8.1 mmol/L) in men at screening.
10. Any exclusion specific to paritaprevir/ritonavir/ombitasvir, dasabuvir or ribavirin.
11. Pregnancy/lactation or male subjects whose female partners are pregnant.
12. Subject has current or past clinical evidence of decompensated liver disease, such as ascites, hepatic encephalopathy, oesophageal varices, and/or any of the following screening laboratory results;

    a. International normalised ration (INR) >1.5; i. Patients with a known inherited blood disorder and INR > 1.5 may be enrolled after discussion with the Principal Investigator b. Serum albumin <3.3 g/dL; c. Serum total bilirubin >1.8 x ULN, unless isolated in subjects with Gilbert's syndrome.
13. Subject shows evidence of significant liver disease in addition to HCV, which may include but is not limited to drug- or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, non-alcoholic steatohepatitis (NASH), or primary biliary cirrhosis.
14. Subject has active malignant disease or history of malignant disease within the past 5 years (except treated basal cell carcinoma).
15. History of chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
16. Poorly controlled diabetes mellitus as evidenced by haemoglobin A1c (HbA1c) ≥8.5%.
17. Positive test at screening for anti-HAV IgM Ab, anti-HBc IgM Ab or HBsAg.
18. Confirmed presence of hepatocellular carcinoma indicated on imaging techniques such as computed tomography (CT) scan or magnetic resonance imaging (MRI) within 3 months prior to screening or on an ultrasound performed at screening (a positive ultrasound result will be confirmed with CT scan or MRI).
19. Subject has history of organ transplant that requires chronic immunosuppression.
20. Corneal, skin, and hair grafts are allowed.
21. History of severe psychiatric disease that in the opinion of the investigator is unstable enough to compromise treatment adherence.
22. Prohibited medications and herbal remedies as detailed in the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with undetectable HCV RNA at 12 weeks post end of treatment (SVR12) | 12 weeks post treatment
  To evaluate the proportion of participants with undetectable HCV RNA 12 weeks post end of treatment (SVR12) following the "3D" regimen with or without ribavirin for 12 weeks in people with chronic HCV genotype 1 infection.

SECONDARY OUTCOMES:
The proportion of participants with undetectable HCV RNA at 2 weeks following the initiation of treatment - week 2 | 2 weeks following the initiation of treatment
  To evaluate the proportion of participants with undetectable HCV RNA after receiving 2 weeks of "3D" regimen with or without ribavirin.
The proportion of participants with undetectable HCV RNA at 4 weeks following the initiation of treatment - week 4 | 4 weeks following the initiation of treatment
  To evaluate the proportion of participants with undetectable HCV RNA after receiving 4 weeks of "3D" regimen with or without ribavirin.
The proportion of participants with undetectable HCV RNA at the end of treatment - week 12 | End of treatment week 12
  To evaluate the proportion of participants with undetectable HCV RNA at the end of treatment after receiving 12 weeks of "3D" regimen with or without ribavirin.
The proportion of participants with undetectable HCV RNA at 24 weeks post end of treatment (SVR24) | 24 weeks post treatment
  To evaluate the proportion of participants with undetectable HCV RNA 24 weeks (SVR24) post end of treatment.
Treatment adherence | Baseline to week 12
  To evaluate the proportion of participants adherent to treatment (both on-treatment adherence and treatment discontinuation).
Association between adherence and response to treatment | Early (0-3 weeks), mid (4-7 weeks), late (8-11 weeks) during treatment
  To evaluate the association between adherence and response to treatment [including an evaluation of the impact of early (0-3 weeks), mid (4-7 weeks) and late (8-11 weeks) missed doses on response to treatment]; adherence will be measured via a self report questionnaire and pill count via return of the weekly blister packs. The impact of the number and timing of the missed pills will be evaluated.
Safety and tolerability (number and type of adverse events and serious adverse events) | Baseline to week 24 (SVR24)
  To evaluate the number and type of adverse events and serious adverse
Change in injecting drug use and injecting risk behaviour | Baseline to week 12
  To evaluate the change in injecting drug use and injecting risk behaviours during and following treatment. Change in injecting drug use and injecting risk behaviour will be measured via a self report behavioural questionnaire completed by participants at baseline, week 4 during treatment, week 8 during treatment and end of treatment.
Change in mental health | Baseline to week 12
  To evaluate the change in mental health during treatment. Change in mental health will be measured by self report mental health questionnaire (Kessler10) at baseline, week 4 during treatment and end of treatment.
Change in health-related quality of life Questionnaire | Baseline to week 12
  To evaluate the change in health-related quality of life during treatment. Change in health-related quality of life will be measured by self report questionnaire (EQ-5D) at baseline, week 4 during treatment and end of treatment.
Impact of mixed HCV infection on treatment response | Baseline to SVR12
  To evaluate the rate of mixed HCV infection at baseline and among those with treatment non-response
Change in opioid substitution therapy | Baseline to week 12
  To evaluate the change in OST during treatment (dose and any discontinuation)
HCV reinfection rate | Week 108
  To evaluate the rate of HCV reinfection during and following treatment
Emergence of viral resistance-associated variants (RAVs) | Baseline to week 12
  To evaluate the emergence of viral resistance-associated variants (RAVs). HCV sequencing will be performed on the baseline EDTA plasma samples of all participants at baseline to detect any baseline RAVs and will be preformed on the EDTA plasma samples of the participants who experienced virological failure to detect the emergence of RAVs.
Utility of HCV core antigen testing as a simple method for HCV monitoring | Week 108
  To evaluate the utility of HCV core antigen testing as a simple method for HCV monitoring including treatment response. HCV RNA will be measured using the HCV core antigen test and then compared to HCV RNA levels measured using standard methods (EDTA plasma samples and Roche TaqMan).

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Dore, MBBS, PhD, Principal Investigator — Kirby Institute
Locations (1):
- The Kirby Institute, University of New South Wales Australia, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cunningham EB, Hajarizadeh B, Amin J, Hellard M, Bruneau J, Feld JJ, Cooper C, Powis J, Litwin AH, Marks P, Dalgard O, Conway B, Moriggia A, Stedman C, Read P, Bruggmann P, Lacombe K, Dunlop A, Applegate TL, Matthews GV, Fraser C, Dore GJ, Grebely J. Reinfection Following Successful Direct-acting Antiviral Therapy for Hepatitis C Virus Infection Among People Who Inject Drugs. Clin Infect Dis. 2021 Apr 26;72(8):1392-1400. doi: 10.1093/cid/ciaa253. PMID 32166305
- [Derived] Artenie AA, Cunningham EB, Dore GJ, Conway B, Dalgard O, Powis J, Bruggmann P, Hellard M, Cooper C, Read P, Feld JJ, Hajarizadeh B, Amin J, Lacombe K, Stedman C, Litwin AH, Marks P, Matthews GV, Quiene S, Erratt A, Bruneau J, Grebely J. Patterns of Drug and Alcohol Use and Injection Equipment Sharing Among People With Recent Injecting Drug Use or Receiving Opioid Agonist Treatment During and Following Hepatitis C Virus Treatment With Direct-acting Antiviral Therapies: An International Study. Clin Infect Dis. 2020 May 23;70(11):2369-2376. doi: 10.1093/cid/ciz633. PMID 31300820